CLINICAL TRIAL: NCT04108403
Title: Mechanisms of Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201902417
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Healthy; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked to the type of instructional set received during the intervention. However, participants will be notified of this upon completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pain Inducing Massage and Positive Expectation Instructions (Experimental): A myofascial trigger point will be assessed in the trapezius muscle and massage applied to this area of the neck. Participants in this arm will receive a positive expectation instructional set followed by a moderately painful massage (pain = 50/100). Massage will be applied for one minute, four times with assessment of pressure pain threshold at the foot between each interval.
  Interventions: Other: Pain Inducing Massage; Other: Positive Expectation Instructional Set
- Pain Inducing Massage and Negative Expectation Instructions (Active Comparator): A myofascial trigger point will be assessed in the trapezius muscle and massage applied to this area of the neck. Participants in this arm will receive a negative expectation instructional set followed by a moderately painful massage (pain = 50/100). Massage will be applied for one minute, four times with assessment of pressure pain threshold at the foot between each interval.
  Interventions: Other: Pain Inducing Massage; Other: Negative Expectation Instructional Set
- Pain Free Massage and Positive Expectation Instructions (Active Comparator): A myofascial trigger point will be assessed in the trapezius muscle and massage applied to this area of the neck. Participants in this arm will receive a positive expectation instructional set followed by a pain free massage (pain = 0/100). Massage will be applied for one minute, four times with assessment of pressure pain threshold at the foot between each interval.
  Interventions: Other: Pain Free Massage; Other: Positive Expectation Instructional Set
- Pain Free Massage and Negative Expectation Instructions (Active Comparator): A myofascial trigger point will be assessed in the trapezius muscle and massage applied to this area of the neck. Participants in this arm will receive a negative expectation instructional set followed by a pain free massage (pain = 0/100). Massage will be applied for one minute, four times with assessment of pressure pain threshold at the foot between each interval.
  Interventions: Other: Pain Free Massage; Other: Negative Expectation Instructional Set

INTERVENTIONS:
Other: Pain Inducing Massage — A pain inducing massage (pain intensity = 50/100) will be applied for 60 seconds, 4 times.
  Arms: Pain Inducing Massage and Negative Expectation Instructions; Pain Inducing Massage and Positive Expectation Instructions
Other: Pain Free Massage — A pain free massage (pain intensity = 0/100) will be applied for 60 seconds, 4 times.
  Arms: Pain Free Massage and Negative Expectation Instructions; Pain Free Massage and Positive Expectation Instructions
Other: Positive Expectation Instructional Set — Participants will be instructed that the massage is effective for some people with neck pain.
  Arms: Pain Free Massage and Positive Expectation Instructions; Pain Inducing Massage and Positive Expectation Instructions
Other: Negative Expectation Instructional Set — Participants will be instructed that the massage is ineffective for some people with neck pain.
  Arms: Pain Free Massage and Negative Expectation Instructions; Pain Inducing Massage and Negative Expectation Instructions

SUMMARY:
The investigators have previously found moderately painful massage produces comparable changes in pain sensitivity as a conditioned pain modulation paradigm in healthy participants suggesting shared underlying mechanisms. The researchers aim to extend these findings by understanding the influence of expectation on these findings.

DETAILED DESCRIPTION:
Massage is a muscle biased intervention individuals seek for pain alleviation; however, the mechanisms of massage are not well established. In this study, the investigators aim to determine the effect of expectations on massage related hypoalgesia. Individuals meeting eligibility criteria and agreeing to participate will attend one session that lasts approximately one hour. A myofascial trigger point (taut band of muscle tissue) will be assessed on the neck of the participant. Next, a baseline assessment of pressure pain threshold will be performed followed by random assignment to one of four study arms.

ELIGIBILITY:
Inclusion Criteria:

* Pain Free

Exclusion Criteria:

* non-English speaking
* systemic medical condition known to affect sensation (i.e. diabetes)
* regular use of prescription pain medication to manage pain
* current or history of chronic pain condition
* currently using blood thinning medication
* any blood clotting disorder such as hemophilia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | 1 hour
  A computerized pressure algometer with a 1cm diameter rubber tip will be applied to the web space of the non-dominant foot. Participants are instructed to say "stop" so the stimulus can be terminated when the sensation first transitions from pressure to pain (threshold).

CONTACTS AND LOCATIONS:
Overall Officials: Joel Bialosky, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson AT, Bishop MD, Beneciuk JM, Tilley HE, Riley JL 3rd, Cruz-Almeida Y, Bialosky JE. Expectations affect pain sensitivity changes during massage. J Man Manip Ther. 2023 Apr;31(2):84-92. doi: 10.1080/10669817.2022.2118449. Epub 2022 Sep 7. PMID 36069038